CLINICAL TRIAL: NCT00311987
Title: A Randomized, Double-Blind Placebo-Controlled Study of 3,5-diiodothyropropionic Acid (DITPA) in Combination With Standard Therapy to Attain NCEP ATP III Goal for LDL Cholesterol in Hypercholesterolemic Patients
Brief Title: Study of 3,5-Diiodothyropropionic Acid (DITPA) in Hypercholesterolemic Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Curtailment of funding by sponsor
Sponsor: Johns Hopkins University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00001376
Record Dates: First submitted 2006-04-05; First posted 2006-04-07 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2006-04

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolemia; Thyroid hormone; Diiodothyropropionic acid; Therapy
MeSH Terms: conditions — Hypercholesterolemia | interventions — 3,5-diiodothyropropionic acid; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 3,5-Diiodothyropropionic acid (DITPA) therapy

SUMMARY:
The natural thyroid hormones, thyroxine (T4) and triiodothyronine (T3), are known to have a cholesterol-lowering effect. Their pharmacologic use for this purpose is limited, however, by their actions on other organs, including the heart, bone, and brain, where there can be side effects of excessive thyroid hormone action. 3,5-diiodothyropropionic acid (DITPA) is a thyroid hormone analog with relative selectivity for a form of the thyroid hormone receptor expressed in the liver, where it regulates several aspects of lipid metabolism, including the clearance of low-density lipoprotein (LDL) cholesterol.

This study is designed to determine whether DITPA is safe and effective in achieving LDL cholesterol levels that are consistent with the National Cholesterol Education Program Adult Treatment Panel III (NCEP ATP III) guidelines in patients who have not achieved those levels on conventional therapy, due to drug-resistant disease, drug intolerance, or both.

This is a single-center, randomized, double-blind, placebo-controlled study. Following a 4-week Pre-Randomization Phase with dietary counseling and a 2-week placebo run-in, eligible patients will be randomized (1:1:1) to receive DITPA (90 mg/day, 180 mg/day), or placebo for a total treatment duration of 12 weeks.

Sixty (60) patients will be randomized to 1 of 3 treatment groups in a 1:1:1 ratio (i.e., 20 patients per treatment group):

* DITPA at 90 mg/day (45 mg twice a day [BID] taken orally)
* DITPA at 180 mg/day (90 mg BID taken orally)
* Placebo (BID taken orally)

Those patients randomized to receive DITPA at 90 mg/day will receive 45 mg/day for the first 2 weeks, followed by 90 mg/day for 10 weeks.

Those patients randomized to receive DITPA at 180 mg/day will receive 45 mg/day for the first 2 weeks, followed by 90 mg/day for the next 2 weeks, and then 180 mg/day for 8 weeks.

DETAILED DESCRIPTION:
INTRODUCTION

BACKGROUND: In recent years, the need to achieve increasingly ambitious therapeutic goals for dyslipidemias has prompted the search for more potent pharmacological agents to lower circulating atherogenic lipoprotein concentrations and enhance reverse cholesterol transport (RCT). While mounting evidence supports the use of 3-hydroxy-3-methylglutaryl coenzyme reductase inhibitors (or statins) as the main stay of therapy for patients requiring lipid modification therapy, many patients remain under-treated or do not achieve the National Cholesterol Education Program (NCEP) recommended goals.1-5 Recognizing new and emerging data, NCEP III recently updated its guidelines to recognize the potential of a more aggressive low density lipoprotein (LDL) goal of <70 mg/dl in patients at high risk of cardiovascular events.3 The Treating to New Targets (TNT) study showed that even in patients with stable coronary artery disease, a goal that is lower than currently recommended, <80 mg/dl, may be desirable in further reducing and/or preventing recurrent cardiovascular events.6 More than 40% of all Americans have LDL levels of 130 mg/dl or higher, and 13 million Americans have coronary artery disease that may benefit from lipid modification therapy. In these individuals, to achieve the optimal LDL goal and to treat other associated lipid abnormalities, including low HDL cholesterol and/or high triglycerides, many patients will likely require combination therapy.3, 7-13 Among the novel therapeutic agents investigated have been selective thyroid hormone analogues. Such agents hold the promise of harnessing the cholesterol-lowering properties of the naturally occurring thyroid hormones, triiodothyronine (T3) and thyroxine (T4), but with greater receptor isoform and tissue specificity that should result in an improved safety profile.14, 15 Unlike statins, thyroid hormones and their analogues, in addition to cholesterol and LDL-lowering effects, may favorably lower lipoprotein (a) (Lp(a)) and triglyceride levels.15-22 Also, because of potential thyroid hormone-mediated genomic and non-genomic effects on the heart, certain populations, such as those with congestive heart failure, may derive dual benefits from use of such thyromimetic treatment.15, 22, 23 1.1.1 Effects of Thyroid Hormone on Lipid Metabolism Dyslipidemia has long been associated with disorders of thyroid metabolism (i.e., hypothyroidism) and to be potentially reversible by thyroid hormone therapy.17, 18, 21 Early autopsy series demonstrated more severe atherosclerosis in individuals with premorbid hypothyroidism.24, 25 In studies of how thyroid hormone status affected radiolabeled lipoprotein kinetics, LDL was found to be cleared less rapidly in hypothyroid animals and man.26 Subsequently, hepatic LDL receptor number27 and mRNA expression28 were shown to be lower in hypothyroid animals. More recently, characterization of the LDL receptor gene promoter has revealed the presence of functionally important T3 regulatory elements.29 In addition to lowering total and LDL cholesterol concentrations in treated hypothyroid patients, thyroid hormone therapy has been shown in some studies to have a favorable impact on particularly atherogenic lipoproteins, including Lp(a)30 and small dense and oxidizable LDL subfractions.31, 32 Finally, thyroid hormone replacement therapy has been shown to decrease apoB100 lipoprotein synthesis with a resulting decrease in Very Low Density Lipoprotein (VLDL) production and hepatic triglyceride production.33 There is now also considerable evidence that thyroid hormone receptor agonists can directly or indirectly affect reverse cholesterol transport, the process by which cholesterol is transported from peripheral cells, including cholesterol-laden endothelial cells in the initial stage of atherosclerosis, to the liver for conversion to bile acids. First, thyroid hormone affects the activity of apoA 1 lipoprotein,34 which plays several critical roles in RCT-generating HDL that transports cholesterol from peripheral tissues to the liver, as both the principal protein constituent of HDL and an activator of lecithin-cholesterol acyltransferase (LCAT), which esterifies cholesterol on the surface of pre-β-HDL. ApoA-I also stabilizes and increases the level of ATP-binding cassette A1 protein (ABCA1), which, in turn, promotes efflux of cholesterol and phospholipids to nascent HDL-particles. Thyroid hormone increases apoA-I gene expression in liver and intestine, in part through a 5' flanking thyroid hormone response element.35, 36 Thyroid hormone has also recently been shown to increased the scavenger class B type I receptor (SR-BI), another regulator of serum HDL concentrations and cholesterol flux, in livers of mice treated with either T3 or GC-1 (a thyroid hormone receptor modulator).37 Finally, thyroid hormones are also known to increase activity of cholesterol 7α-hydroxylase (CYP-7A1)38 which catalyzes the rate-limiting step in bile acid synthesis; in contrast, HMG-CoA reductase inhibitors have the opposite effect. This thyroid hormone-induced increase in CYP-7A1 would be expected to increase bile acid and cholesterol excretion, as has been observed in hyperthyroidism.39 1.1.2 Previous Clinical Research Previous studies have investigated the therapeutic potential of thyromimetic compounds in lipid modification and heart failure.14,15,40 Early clinical investigation focused on dextrothyroxine (D-T4), a D-isomer of thyroxine, which was thought to have similar actions, but produce less tachycardia and myocardial oxygen consumption.40, 41 Although DT4 was commonly used as a cholesterol lowering drug in the 1970s,42 it is no longer used in clinical practice. The therapeutic effects of DT4 were evaluated in the Coronary Drug Project (CDP).

The Coronary Drug Project was initiated in 1965, primarily to answer the prevailing question about the safety and efficacy of long term use of various cholesterol lowering agents in patients with coronary artery disease. The Coronary Drug Project was a randomized, double-blind, placebo-controlled study, conducted between 1966 and 1975. It was designed to evaluate the efficacy and safety of five lipid-modifying drugs in 8,341 men, with a history of prior myocardial infarction (MI). Niacin, clofibrate, dextrothyroxine, and two estrogen regimens were evaluated in the study along with a placebo arm.43, 44 DT4 was administered at 6.0 mg /day. The primary endpoint was overall mortality at 5 years. After a mean follow-up of 36 months, because of a nonsignificant trend toward higher mortality in the DT4 arm compared with placebo, the DT4 arm was discontinued.

As acknowledged by the original investigators, the observed DT4-placebo difference in overall mortality is not statistically significant as judged by the statistical methods utilized in this study.44 Nevertheless, given the mortality trend and the low probability of eventual benefits, a decision was made to discontinue the DT4 arm. In discontinuing the DT4 arm, the study leadership recognized that the findings of the CDP left open the possibility that dextrothyroxine may be efficacious for a limited group of carefully selected myocardial infarction (MI) patients and for persons free of clinical CHD. 44 The net effect of DT4 on serum lipids (the observed fall corrected for the concomitant rise for the placebo group) was a sustained significant fall from baseline levels. The decrease was approximately 12% in serum cholesterol levels and 15-20% in fasting serum triglyceride levels.44 Following the study, it was revealed that the DT4 dispensed in the study contained less than 0.5% of levothyroxine (approximately 30 µg of levothyroxine).44 Interestingly, it was later found that contamination of levothyroxine commercial preparations varied from lot to lot (from 0.5% to 2.3%).45 Also, this "DT4" formulation had other significant thyromimetic effects, leading to TSH suppression that may have become clinically relevant with prolonged use.47 Suboptimal dosing and thyrotoxic effects due to drug contamination may explain why more than 40% of the DT4 patients required a dose reduction.44 1.1.3 DITPA DITPA (3,5-diiodothyropropionic acid) is an analogue of naturally occurring thyroid hormone (T3) that has been specifically designed to improve cardiac performance with a lower potential for tachycardia.22, 40, 46 DITPA binds to the same thyroid hormone receptors α and β as T3 but with less affinity.41 In pre-clinical animal post-infarction models, DITPA improved calcium handling, promoted angiogenesis, and attenuated abnormal left ventricular remodeling.47-53 In a rat model of CHF, DITPA demonstrated increased cardiac output with increases in left ventricular dp/dt, comparable to effects seen with T4, but with significantly less tachycardia. In addition, there were increases in α-myosin heavy chain (MHC) RNA gene expression induced by DITPA treatment.41 When evaluated in combination with captopril, DITPA improved both cardiac output and dp/dt as well as increased the rate of LV relaxation when compared with captopril alone.54 In a rabbit post-infarction model, DITPA decreased left ventricular end diastolic pressure and increased positive and negative dp/dt without changes in heart rate or left ventricular systolic pressure.43 In the same model, use of DITPA prevented abnormal SERCA transport and abnormal contractile function associated with myocardial infarction.42, 44 Recently DITPA was also noted to improve endothelial function following myocardial infarction, an action mediated through nitric oxide.55 The objective of the present study is to evaluate the feasibility of DITPA, a thyroid hormone analogue, as a potential lipid modification agent.

KNOWN AND POTENTIAL TOXICITIES: Since DITPA is a thyroid hormone analogue with thyromimetic actions, safety and side effect profiles may be similar to those observed with thyroid hormones T3 and T4 preparations (e.g., liothyronine and levothyroxine). Although excess thyromimetic action is a theoretical side effect, it is also possible that tissue-specific hypothyroidism might result if the drug fails to have sufficient thyromimetic activity in a particular tissue. Due to pituitary effects of DITPA, a secondary lowering of TSH may result, which in turn may lead to decreased endogenous production of T4. The potential effects of such theoretical biochemical changes are unknown. Thus, DITPA safety will be diligently monitored throughout the study through multiple examinations, symptom scales, and laboratory evaluations.

Based on the known effects of thyrotoxicosis and hypothyroidism, and the side effects of T3 and T4 preparations, potential side effects of DITPA may include:

1. Cardiovascular: palpitations, tachycardia, arrhythmias, increased pulse and blood pressure, heart failure, angina, myocardial infarction, cardiac arrest
2. Central nervous system: headache, hyperactivity, nervousness, anxiety, irritability, emotional lability, insomnia
3. Dermatologic: hair loss, warm moist or dry skin, flushing
4. Endocrine: decreased bone mineral density, gynecomastia
5. Gastrointestinal: diarrhea or constipation, vomiting, abdominal cramps, elevations in liver function tests
6. General symptoms: fatigue, increased appetite, excessive sweating
7. Musculoskeletal: tremors, muscle weakness, proximal myopathy
8. Respiratory: dyspnea
9. Reproductive: menstrual irregularities, impaired fertility
10. Metabolic: weight loss or gain, heat or cold temperature intolerance, fever Please consult the most recent DITPA Investigator's Brochure (IB) including amendments for additional information.

In addition, many drugs are known to affect thyroid hormone pharmacokinetics and metabolism by altering absorption, synthesis, secretion, protein binding, and/or target tissue response, and may also alter the therapeutic response to thyroid hormone preparations such as levothyroxine. In addition, thyroid hormones and thyroid status may have varied effects on the pharmacokinetics and actions of other drugs. A list of drug-thyroidal axis interactions is provided in the prescribing information for marketed agents such as Synthroid® (levothyroxine sodium tablets, USP), Abbott Laboratories and Cytomel® (liothyronine sodium tablets), King Pharmaceuticals, Inc.

STUDY DESCRIPTION

STUDY OBJECTIVES:

Primary Objective

* To evaluate DITPA as a lipid modifying agent in combination with standard therapy in patients with LDL-C levels greater than the NCEP ATP III goals as determined by patient's risk category, in order to achieve NCEP III LDL-C goals (see Appendix C).

Secondary Objectives

* To evaluate the effect of DITPA on other lipid targets: triglyceride, total cholesterol , ratio of total cholesterol to HDL, ratio of LDL to HDL, HDL cholesterol, lipoprotein a (Lp (a)), apolipoprotein A-I, apolipoprotein B100, and LDL subfractions
* To evaluate the effect of DITPA on weight and waist circumference
* To evaluate the effect of DITPA on high sensitive C-reactive protein (hs CRP)
* To evaluate the safety of DITPA in this patient population

STUDY DESIGN: This is a single-center, randomized, double-blind, placebo-controlled study to evaluate hyperlipidemic patients on standard lipid-lowering therapy with LDL-C levels exceeding NCEP ATP III goals. Following a 4-week Pre-Randomization Phase with dietary counseling and a 2-week placebo run-in, eligible patients will be randomized (1:1:1) to receive DITPA (90 mg/day, 180 mg/day), or Placebo for a total treatment duration of 12 weeks.

Sixty 60 patients will be randomized to 1 of 3 treatment groups in a 1:1:1 ratio (i.e., 20 patients per treatment group):

* DITPA at 90 mg/day (45 mg BID taken orally)
* DITPA at 180 mg/day (90 mg BID taken orally)
* Placebo (BID taken orally)

Those patients randomized to receive DITPA at 90 mg/day will receive 45 mg/day for the first 2 weeks, followed by 90 mg/day for 10 weeks.

Those patients randomized to receive DITPA at 180 mg/day will receive 45 mg/day for the first 2 weeks, followed by 90 mg/day for next 2 weeks, and then 180 mg/day for 8 weeks.

Q1, Q2 = first and second qualifying LDL cholesterol values using Friedewald's calculation

STUDY DURATION AND NUMBER OF VISITS: The study will consist of a Screening Phase with ATP III diet counseling, a Pre-Randomization Phase that will consist of dietary counseling plus a 2-week Placebo Run-In Period, and a 12-week Treatment Phase. Patients will be seen 28 days after the End of Treatment Visit. The total duration on study will be approximately 20 weeks.

Patients will be seen for approximately 9 visits: Screening visit, 2 Pre-Randomization visits (Q1 and Q2), a Baseline/Week 0 visit, Week 2, 4, 8, 12/ End of Treatment visits, and a Week 16/Follow-up visit.

STUDY DRUG

STUDY DRUG TREATMENTS TO BE ADMINISTERED: DITPA Capsules 3,5-Diiodothyropropionic acid, or DITPA, is the active pharmaceutical ingredient (API). The chemical structure of DITPA is shown below: Molecular Formula: C15H12I2O4 Molecular Weight: 510.1 Chemical Name: 3,5-diiodothyropropionic acid

DOSING INFORMATION: Patients should be instructed to take 1 capsule in the morning 30 minutes before breakfast, and 1 capsule in the evening 30 minutes before the evening meal. The 2 doses should be taken approximately 10-12 hours apart. Capsules should be taken by mouth with a full glass of water. Patients should be instructed not to crush, break, or chew the capsules, and to swallow the capsules whole.

BLINDING: Treatment assignments and administration will be double-blinded. All patients will receive medication cards containing study drug capsules (active and/or placebo). The 45 mg, 90 mg, and placebo capsules will appear identical and the dose will be unidentifiable.

STUDY SUBJECTS

STUDY POPULATION: The study population consists of patients who have LDL-C levels greater than NCEP III ATP goals as determined by patient's risk category despite standard lipid modification therapy.

CRITERIA TO ENTER STUDY (PRE-RANDOMIZATION PHASE)

Pre-Randomization Criteria:

Patients are eligible for study entry based on the following criteria:

1. Male or female greater than or equal to 18 years of age
2. Females must not be pregnant or lactating. Females of childbearing potential and males must use a reliable means of contraception
3. LDL-C level greater than the NCEP goals as determined by patients' risk category according to NCEP ATP III criteria
4. Risk category for coronary heart disease and coronary heart disease equivalent with LDL goal of <100 mg/dL
5. Baseline lipid criteria: LDL-C = 100 to160 mg/dL and Triglyceride level = 100 to 500 mg/dL
6. Normal Thyroid Function Tests (total T3, total T4, and TSH)
7. Hemoglobin A1C <8.5 % on a stable oral hypoglycemic or insulin regimen
8. On stable lipid modification pharmacotherapy (including a statin) for at least 2 weeks prior to study entry. Patients must be on at least half maximal doses of statins (as assessed by the Investigator), or be intolerant to statins such that the doses are not achievable.
9. Able to give informed consent

Pre-randomization Exclusion Criteria:

Patients will not be eligible for the study based on the following criteria:

1. History of thyroid disorders of any form within 24 weeks prior to study entry
2. Active liver disease and/or liver transaminases greater than 1.5 X upper limit of normal
3. Active myocarditis, hypertrophic cardiomyopathy, uncorrected primary valvular disease, restrictive cardiomyopathy, uncorrected congenital heart disease, or constrictive pericarditis
4. Myocardial infarction, unstable ischemic heart disease, stroke, or coronary revascularization procedure within 24 weeks prior to study entry
5. Moderate or severe symptomatic congestive heart failure (New York Heart Association class III and IV)
6. Drug or alcohol dependence, or other conditions which may affect study compliance
7. Renal insufficiency (serum creatinine > 2 mg/dL)
8. Subjects taking other hormonal therapies (other than oral contraceptive agents and postmenopausal hormone replacement therapy) e.g., glucocorticoids, androgens, or growth hormones
9. Use of thyroid supplements (levothyroxine, liothyronine, etc.) or any preparation containing thyromimetic agents within 24 weeks prior to study entry
10. History of coagulopathy or use of anticoagulants such as warfarin
11. Unstable endocrine/metabolic syndrome that may affect lipid metabolism
12. History of atrial or ventricular arrhythmia
13. Diagnosis of other non-cardiac underlying medical conditions expected to impact their mortality within 24 weeks after randomization

CRITERIA FOR RANDOMIZATION

Randomization Inclusion Criteria:

Patients are eligible for randomization based on the following criteria:

1. LDL-C level greater than the NCEP goals as determined by patients' risk category according to NCEP ATP III criteria
2. Risk category for coronary heart disease and coronary heart disease equivalent with LDL goal of <100 mg/dL
3. Baseline lipid criteria: LDL-C = 100 to160 mg/dL (as calculated from Q1 and Q2 lipid results) and Triglyceride level = 100 to 500 mg/dL
4. If on anti-hypertensive therapy, therapy must be stable for at least 4 weeks prior to randomization
5. Stable lipid modification pharmacotherapy for at least 6 weeks prior to randomization
6. Compliance with medication dosing instructions during the single-blind placebo run -in period is 80% to 120% as measured by pill counting.

Randomization Exclusion Criteria:

Patients will not be eligible for randomization based on the following criteria:

1. Significant changes in clinical status from the Screening Visit which would preclude the patient from being an appropriate candidate.

   STUDY PROCEDURES: Refer to Appendix A: Schedule of Events for the Sequence and Timing of Study Procedures. While every effort must be made to adhere to the schedule, there will be a ± 5 day window for each study visit. All visits are in reference to the date of randomization.

   SCREENING (VISIT 1):

   A signed informed consent must be obtained prior to any study-specific procedures. The following procedures are to be completed at the Screening Visit (4 to 8 weeks prior to randomization):
   * Review list of inclusion/exclusion pre-randomization criteria
   * Collect laboratory samples:

     * Hematology/chemistry
     * Urine sample
     * Pregnancy test
     * Thyroid function tests
     * Fasting lipid panel
     * Future tests may include lipoprotein (a), NMR lipoprotein subfraction analysis, homocysteine, inflammatory markers (PAI-1, selectins, interleukins, myeloperoxidase, matrix metalloproteinases) and markers for metabolism (leptin and adiponectin)
   * Dietary counseling (ATP III)

   PRE-RANDOMIZATION VISIT (Q1 - VISIT 2):
   * Collect laboratory samples: Fasting lipid panel (first qualifying LDL-C (Q1))
   * Dietary counseling (ATP III)

   PLACEBO RUN-IN VISIT (Q2 - VISIT 3):
   * Collect laboratory samples:

     * Fasting lipid panel (second qualifying LDL-C (Q2))
     * PT/INR
     * Future tests may include lipoprotein (a), NMR lipoprotein subfraction analysis, homocysteine, inflammatory markers (PAI-1, selectins, interleukins, myeloperoxidase, matrix metalloproteinases) and markers for metabolism (leptin and adiponectin)
     * Assess patient for qualifying mean calculated LDL-C
   * Dietary counseling (ATP III)
   * Dispense placebo 2-week medication card

   BASELINE (VISIT 4):

   Once the patient is deemed eligible, the following baseline procedures should be completed within 7 days prior to randomization:
   * Assess patient drug compliance (placebo run-in)
   * Review list of inclusion/exclusion randomization criteria
   * Obtain a patient randomization number and kit number (within 2 days prior to study drug administration)
   * Review medical and medication history
   * Physical examination, vital signs, weight, height, eye examination, waist measurement
   * DEXA scan for body fat composition and bone mineral density
   * Thyroid symptom assessments: Hyperthyroid Symptom Scale, Modified Billewicz Index for Hypothyroidism, and Hypothyroid Symptom Scale
   * Echocardiogram
   * Electrocardiogram (ECG)
   * Collect laboratory samples:

     * Hematology/chemistry
     * Urinalysis
     * hsCRP
     * Serum bone markers (osteocalcin, N-telopeptides)
     * Pregnancy test
     * Thyroid function tests
     * Fasting lipid panel
     * Future tests may include lipoprotein (a), NMR lipoprotein subfraction analysis, homocysteine, inflammatory markers (PAI-1, selectins, interleukins, myeloperoxidase, matrix metalloproteinases) and markers for metabolism (leptin and adiponectin)
     * PT/INR
     * DITPA concentration
   * Pre-randomization adverse events and concomitant medications

   TREATMENT PERIOD (VISIT 5):
   * Obtain a new kit number
   * Physical examination, vital signs, weight, eye examination, waist measurements
   * Thyroid symptom assessments: Hyperthyroid Symptom Scale, Modified Billewicz Index for Hypothyroidism, and Hypothyroid Symptom Scale
   * Adverse events and concomitant medications
   * Collect laboratory samples:

     * Thyroid function tests
     * Fasting lipid panel
     * Future tests may include lipoprotein (a), NMR lipoprotein subfraction analysis, homocysteine, inflammatory markers (PAI-1, selectins, interleukins, myeloperoxidase, matrix metalloproteinases) and markers for metabolism (leptin and adiponectin)
     * DITPA concentration
   * Dispense study drug and assess study drug compliance

   TREATMENT PERIOD (VISIT 6):
   * Obtain a new kit number
   * Physical examination, vital signs, weight, eye examination, waist measurement
   * Thyroid symptom assessments: Hyperthyroid Symptom Scale, Modified Billewicz Index for Hypothyroidism, and Hypothyroid Symptom Scale
   * ECG
   * Adverse events and concomitant medications
   * Collect laboratory samples:

     * Hematology/chemistry
     * Urinalysis
     * Pregnancy test
     * Thyroid function tests
     * Fasting lipid panel
     * Future tests may include lipoprotein (a), NMR lipoprotein subfraction analysis, homocysteine, inflammatory markers (PAI-1, selectins, interleukins, myeloperoxidase, matrix metalloproteinases) and markers for metabolism (leptin and adiponectin)
     * PT/INR
     * DITPA concentration
   * Dispense study drug and assess study drug compliance

   TREATMENT PERIOD (VISIT 7):
   * Obtain a new kit number
   * Physical examination, vital signs, weight, eye examination, waist measurement
   * Adverse events and concomitant medications
   * Collect laboratory samples:

     * Hematology/chemistry

     * Urinalysis
     * Pregnancy test
     * Fasting lipid profile
     * DITPA concentration
   * Dispense study drug and assess study drug compliance

   END OF TREATMENT VISIT (VISIT 8): Study patients who have completed 12 weeks of treatment, or who have discontinued early (prior to Week 12) will be evaluated at the End of Treatment visit. If evaluations were performed within 1 week of discontinuation, they do not need to be repeated, unless follow-up for safety concerns is needed.

   The following Week 12/Visit 8 study procedures should be completed:
   * Physical examination, vital signs, weight, eye examination, waist measurement
   * DEXA scan for body fat composition and bone mineral density
   * Thyroid symptom assessments: Hyperthyroid Symptom Scale, Modified Billewicz Index for Hypothyroidism, and Hypothyroid Symptom Scale
   * Echocardiogram
   * ECG
   * Adverse events and concomitant medications
   * Collect laboratory samples:

     * Hematology/chemistry

     * Urinalysis

     * HsCRP

     * Serum bone markers

     * Pregnancy test

     * Thyroid function tests

     * Fasting lipid panel

     * Future tests may include lipoprotein (a), NMR lipoprotein subfraction analysis, homocysteine, inflammatory markers (PAI-1, selectins, interleukins, myeloperoxidase, matrix metalloproteinases) and markers for metabolism (leptin and adiponectin)

     * PT/INR
   * Study drug compliance

   FOLLOW-UP VISIT (VISIT 9):

   Study patients will be seen 28 days after the End of Treatment visit. The following procedures should be completed during this visit:

   - Physical examination, vital signs, weight, eye examination, waist measurement

   - Assess adverse events and concomitant medications

   - Collect laboratory samples:

   * Hematology/chemistry

   * Urinalysis
   * Pregnancy test
   * Thyroid function tests
   * Fasting lipid profile

   UNSCHEDULED VISITS: Study patients should be evaluated and managed following best medical practice with particular attention paid to patient safety, assessment of potential treatment-related adverse events, and changes in clinical status.

   EVALUATIONS: Study patients will be closely monitored throughout the study for safety and clinical response. The results of all safety and efficacy evaluations must be recorded in the CRF and in the source documents.

   DESCRIPTION OF EVALUATIONS AND STUDY-SPECIFIC PROCEDURES

   Informed Consent: Patients must give written informed consent, after the nature of the study has been fully explained, in order to participate in this study. No study-specific procedures may be performed before written informed consent is obtained.

   Randomization of Patients: Patients who sign an Informed Consent Form (ICF), complete all screening evaluations, pre-randomization (qualification) evaluations, and meet all entry criteria, will be eligible for randomization, and enrollment into the study. Randomization should occur within 2 days prior to study drug administration. All patients will be randomized in a 1:1:1 fashion to 1 of 3 treatment groups in order to reduce selection bias. All randomization will be managed centrally, by the GCRC.

   Medical and Medication History: A complete record of the patient's medical history, other medical conditions, and concomitant medications (including current lipid modification agents) will be obtained and recorded in the medical chart and CRF.

   Physical Examination, Vital Signs, and Weight: Patients will be seen by an Investigator for a complete physical examination, vital signs (temperature, systolic and diastolic blood pressure, pulse, and respiration rate), waist measurement and weight. Height will be measured at baseline only. The eye examination, including a funduscopic exam and measurement of visual acuity, will be conducted at the Baseline Visit and End of Treatment Visit only.

   Thyroid Symptom Assessment: Three clinical symptom scales (Hyperthyroid Symptom Scale,60 Modified Billewicz Index for Hypothyroidism,61, 62 and the Hypothyroid Symptom Scale) will be used to assess and document potential thyroid-related symptoms. See attachment B for details. The hypothyroid scale is a patient self-assessment and will be completed by the patient at the beginning of the visit. The hyperthyroid scale and modified Billewicz will be completed by the Investigator or designee. The same scales are currently in use in the ongoing DITPA studies.

   Echocardiogram: An echocardiogram will be performed at Baseline and Visit 8/End of Treatment Visit for safety monitoring. The echocardiograms will be interpreted by a designated study cardiologist for safety and efficacy, in a blinded fashion.

   Electrocardiogram (ECG): An electrocardiogram should be performed at the specified visits.

   DEXA Scan: Dual Energy X-ray Absorptiometry, or DEXA scanning, will be used to measure bone mineral density and body fat composition.

   Laboratory Evaluations:

   The following laboratory testing will be performed according to the schedule in Appendix A:

   Hematology Hemoglobin, Hemoglobin A1C, Hematocrit, RBC, MCV, MCH, RBC Morphology, WBC with differential, and platelets Chemistry Total Bilirubin, Alkaline Phosphatase, ALT (SGPT), AST (SGOT), GGT, LDH, Urea Nitrogen (BUN), Creatinine, Creatinine Kinase, fasting Glucose, Serum Calcium, Phosphorus, Total Protein, Albumin, Sodium, Uric Acid, Potassium, HCO3, Amylase, and Chloride Urinalysis Blood, nitrites, protein, ketones, glucose, pH, and specific gravity Pregnancy test Human chorionic gonadotropin (HCG) assay Thyroid Function Tests Total T3, Total T4, and TSH Fasting Lipid Panel Low-density lipoprotein (LDL) cholesterol, high-density lipoprotein (HDL) cholesterol, triglycerides, and total cholesterol Other lipids and future testing* Lipoprotein (a), apolipoprotein A, apolipoprotein B, lipoprotein subfractions by NMR spectroscopy, homocysteine, selectins, interleukins, PAI-1, myeloperoxidase, matrix metalloproteinases, leptin, adiponectin.

   PT/INR Prothrombin time/international normalized ratio Bone marker* Serum osteocalcin and N-telopeptide Inflammatory markers* High Sensitivity CRP (hs CRP) Analysis for DITPA concentrations* Trough steady state levels of DITPA * Testing of samples for these parameters may be performed at a later time, following initial efficacy analysis

   Fasting: Patients will be instructed to fast at least 12 hours prior to Visits 1, 2, 3, 5, 6, 8, and 9 for the fasting lipid panel blood draws.

   Blood draws for DITPA concentrations: Blood for DITPA concentrations will be drawn at least 6 hours after the preceding dose of study drug. It is recommended that if the patient has a morning appointment, the patient should not take the morning dose until after the blood draw. If the patient has an afternoon appointment, the patient should take the morning dose as usual. The time of the preceding dose should be recorded in source documents and the CRF.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible for study entry based on the following criteria:

1. Males or females greater than or equal to 18 years of age
2. Females must not be pregnant or lactating. Females of childbearing potential and males must use a reliable means of contraception.
3. LDL-C level greater than the NCEP goals, as determined by patients' risk category according to NCEP ATP III criteria
4. Risk category for coronary heart disease and coronary heart disease equivalent with LDL goal of < 100 mg/dL
5. Baseline lipid criteria: LDL-C = 100 to160 mg/dL and triglyceride level = 100 to 500 mg/dL
6. Normal thyroid function tests (total T3, total T4, and thyroid-stimulating hormone [TSH])
7. Hemoglobin A1C < 8.5% on a stable oral hypoglycemic or insulin regimen
8. On stable lipid modification pharmacotherapy (including a statin) for at least 2 weeks prior to study entry. Patients must be on at least half of the maximal doses of statins (as assessed by the Investigator), or be intolerant to statins such that the doses are not achievable.
9. Able to give informed consent

Exclusion Criteria:

Pre-Randomization Exclusion Criteria

Patients will not be eligible for the study based on the following criteria:

1. History of thyroid disorders of any form within 24 weeks prior to study entry
2. Active liver disease and/or liver transaminases greater than 1.5 X upper limit of normal
3. Active myocarditis, hypertrophic cardiomyopathy, uncorrected primary valvular disease, restrictive cardiomyopathy, uncorrected congenital heart disease, or constrictive pericarditis
4. Myocardial infarction, unstable ischemic heart disease, stroke, or coronary revascularization procedure within 24 weeks prior to study entry
5. Moderate or severe symptomatic congestive heart failure (New York Heart Association class III and IV)
6. Drug or alcohol dependence, or other conditions which may affect study compliance
7. Renal insufficiency (serum creatinine > 2 mg/dL)
8. Subjects taking other hormonal therapies (other than oral contraceptive agents and postmenopausal hormone replacement therapy) e.g., glucocorticoids, androgens, or growth hormones
9. Use of thyroid supplements (levothyroxine, liothyronine, etc.) or any preparation containing thyromimetic agents within 24 weeks prior to study entry
10. History of coagulopathy or use of anticoagulants such as warfarin
11. Unstable endocrine/metabolic syndrome that may affect lipid metabolism
12. History of atrial or ventricular arrhythmia
13. Diagnosis of other non-cardiac underlying medical conditions expected to impact mortality within 24 weeks after randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-04; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To evaluate DITPA as a lipid modifying agent in combination with standard therapy in patients with LDL cholesterol (LDL-C) levels greater than the NCEP ATP III goals, as determined by patient's risk category, in order to achieve NCEP III LDL-C goals

SECONDARY OUTCOMES:
To evaluate the effect of DITPA on other lipid targets: triglyceride
total cholesterol
ratio of total cholesterol to high-density lipoprotein (HDL)
ratio of LDL to HDL
HDL cholesterol
lipoprotein a [Lp (a)]
apolipoprotein A-I
apolipoprotein B100
and LDL subfractions
To evaluate the effect of DITPA on weight and waist circumference
To evaluate the effect of DITPA on high sensitivity C-reactive protein (hs CRP)
To evaluate the safety of DITPA in this patient population

CONTACTS AND LOCATIONS:
Overall Officials: Annabelle Rodriguez, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States